CLINICAL TRIAL: NCT03964753
Title: The Effectiveness and Safety of Neoadjuvant Therapy With Nab-paclitaxel and Cisplatin Followed by Surgery Versus Surgery Alone for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant Therapy With Nab-paclitaxel and Cisplatin for Locally Advanced Esophageal Squamous Cell Carcinoma
Acronym: NTNC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, LiuJunFeng, Director of thoracic surgery, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HebeiJLiu
Record Dates: First submitted 2019-05-18; First posted 2019-05-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neo-adjuvant chemotherapy group (Experimental): cisplatin and nab-paclitaxel: Nab-paclitaxel, 125mg/m(2), d1,d8, Cisplatin, 75mg/m(2), d1, 3 week, 2 cycles.
  Surgery:
  4-6weeks after Neo-adjuvant chemotherapy
  Interventions: Drug: Nab-paclitaxel and Cisplatin; Procedure: surgery
- Surgery alone (Active Comparator): Surgery alone
  Interventions: Procedure: surgery

INTERVENTIONS:
Drug: Nab-paclitaxel and Cisplatin — Nab-paclitaxel,125mg/m(2), d1,d8, Cisplatin,75mg/m(2), d1, 3 week, 2 cycles.
  Arms: Neo-adjuvant chemotherapy group
Procedure: surgery — surgery

SUMMARY:
To verify the role of nab-paclitaxel in neoadjuvant therapy for esophageal squamous cell carcinoma, the investigators designed a prospective, randomized, controlled , multicente phase II trial, to investigate the efficacy and safety of nab-paclitaxel combined with cisplatin as neoadjuvant therapy followed by surgery versus surgery alone for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 75 years
* Radiographically, histologically or/and cytologically diagnosed resectable locally advanced middle-lower esophageal squamous cell carcinoma without distant metastasis,cT1N1M0 or T2-3N0-1M0(according to UICC esophageal cancer TNM staging system 8th edition)
* Enhanced CT showed the presence of potentially resectable lesions. Resectability features included no evidence of mediastinal infiltration, No evidence of tracheobronchial fistula or tumor entry into the airway
* Have not previously received systemic antitumor therapy for esophageal squamous cell carcinoma (Including radiotherapy, chemotherapy, targeted therapy, immunotherapy)
* ECOG performance status 0-1
* Expected survival more than 6 months
* No contraindications in the organ function tests before surgery
* The laboratory test meet the following requirements:

Bone marrow function: neutrophils ≥ 1.5×10(9)/L, platelets ≥ 100×10(9)/L, hemoglobin ≥ 90 g/L Liver function：Total bilirubin ≤ 1.5x ULN；AST and ALT) ≤ 2.5x ULN Renal function：Cr ≤ 1.5x ULN，Ccr ≥ 55 ml/min Coagulation function：INR≤1.5×ULN, PT≤1.5ULN, APTT within the normal range

* Female patients of child-bearing age agree to take effective contraceptive measures during the study period and 6 months after reseach completion；Pregnancy tests in serum or urine must be negative 7 days prior to study enrollment；Non-lactating patients；male patients agree to take effective contraceptive measures during the study period and 6 months after reseach completion
* Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver)
* Not participating in other clinical trials 4 weeks before the treatment
* The patient has good compliance with the planned treatment, understands the research process of the study and signs a written informed consent form.

Exclusion Criteria:

* Histological confirmation of esophageal adenocarcinoma
* with distant metastasis, without radical resection (stage IV)
* Ever administrated with other drugs(including TCM drugs) before the recruitment, or no guarantee of progress according to the study requirement after recruitment
* Grade 2 or above peripheral neuropathy or hemorrhage according to NCI CTCAE 4.03
* Combined with severe cardiovascular disease, including hypertension that cannot be controlled by medical treatment(BP≥160/95mmHg), unstable angina, a history of myocardial infarction in the past 6 months,Congestive heart failure>NYHA grade II, severe arrhythmia, pericardial effusion, etc.
* Combined with severe ADH abnormal secretion syndrome, poorly controlled diabetes: more than 40 units of insulin per day need to be continuously administered; or 40 units of insulin per day for continuous use or not used, but fasting blood glucose is still above 14mmol / L, HbA1c above 9.0
* Long-term use of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues for more than 6 months,small doses of warfarin (≤1mg / day) or aspirin (≤100mg / day) for prevention purposes are not included
* Major surgery within 4 weeks prior to enrollment, or surgical wounds have not fully healed
* Operation can not use the stomach instead of esophageal cancer to reconstruct the digestive tract due to previous operation
* Severe infection within 1 week prior to the start of study, requiring intravenous antibiotics, antifungal or antiviral therapy
* Known to be allergic, highly sensitive or intolerable to research-related drugs or excipient
* In the past 5 years, there were other malignant tumors, melanoma skin cancer or ervical carcinoma in situ were excepted
* Any indicator shows chemotherapy and surgery contraindications
* Women who are pregnant or lactating
* The investigator determined that unable to complete the study due to medical, social, or psychological reasons or were unable to sign valid informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
OS | up to 5 years
  Overall survival，From date of randomization until death due to any cause

SECONDARY OUTCOMES:
OS rate | 1 year,3years,5years
  Overall survival rate
DFS rate | 1 year,3years,5years
  Disease free survival rate
R0 resection rate | within 4 weeks following the operation
  R0 resection rate
Down-staging rate | within 6 weeks following the last dose of chemotherapy
  Down-staging rate
Rate of Operative Complications | within 4 weeks following the operation
Rate of Adverse Event | up to 6 weeks after the last dose of chemotherapy
  Incidence of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Jun Feng Liu, Shijiazhuang, Hebei, China